CLINICAL TRIAL: NCT00466518
Title: Sitagliptin Treatment in Patients With Type 2 Diabetes Mellitus After Kidney Transplant
Brief Title: Sitagliptin Treatment in Patients With Type 2 DM After Kidney Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 475-06-FB
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Kidney Transplant; Type 2 Diabetes
Keywords: Kidney transplant; type 2 diabetes; sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Administration of sitagliptin

INTERVENTIONS:
Drug: Administration of sitagliptin — Sitagliptin 100 mg daily for 3 months
  Other Names: Januvia

SUMMARY:
This study is designed to look at the effect sitagliptin has on tacrolimus and sirolimus drug levels in kidney transplant patients. It is also designed to look at the side effects experienced in the transplant population.

DETAILED DESCRIPTION:
Within the last six months, the FDA has approved sitagliptin phosphate as an oral drug that potentiates the effect of native GLP-1 through inhibition of DPP-4. It is approved for treatment of type 2 diabetes in adults as monotherapy or in combination with metformin or a TZD. It has several advantages over extenatide when considering its use in kidney transplant recipients:

1. It is administered orally once a day
2. Nausea occurred at a rate of only 1.4%
3. Its potential of hypoglycemia is low

However, it may not be as potent, in terms of HbA1C with % change in HbA1C<1%. In addition there is not a lot of information on gastric emptying, although this is probably not as severe as exenatide, with fewer symptoms of nausea reported.

We propose to conduct a pilot study for using sitagliptin in patients who have both type 2 diabetes and who have received a kidney transplant. Our objectives are to study the effect of sitagliptin administration on side effect profiles, change in HbA1C, and the percentage of patients who require discontinuation of the drug as a result of major changes in immunosuppressant drug levels. The data will be used as preliminary data for a larger study that attempts to prevent or delay the onset of PTDM in kidney transplant recipients. We anticipate treating patients with both impaired fasting glucose and normoglycemia, given the high frequency of PTDM in the post-kidney transplant population.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Most recent HbA1C 6.5-10%
* 1 year post kidney transplant

Exclusion Criteria:

* Patients treated primarily with insulin for their diabetes
* Kidney allograft not functional at entry or estimated creatinine clearance of <30 ml/min
* Clinical course complicated by persistent nausea
* severe gastroparesis
* Severe recurrent hypoglycemia (>1 hypoglycemic episode requiring the help of another person per week).
* Patients on dialysis therapy
* Unstable renal function in the preceding 3 months
* Serum transaminases >2 times normal at study entry
* Smokers
* Pregnant or planning to become pregnant
* Lactating
* Recipients of multi-organ transplants
* Unstable medical conditions which result in multiple hospitalizations or a severely restricted lifestyle
* Hemoglobin <10.0g/dl
* Use of digoxin
* Patients receiving their primary care outside of UNMC
* Inability to come to follow-up visits as a part of the protocol
* Patients not taking tacrolimus and sarolimus as part of their immunosuppressive therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Changes in pharmacokinetics | 3 months

SECONDARY OUTCOMES:
To determine if there is a change in side effects with the addition of sitagliptin to the post-kidney transplant treatment regime. | 3 months
To determine the effect of sitagliptin on glucose lowering over 3 months as measured by the change in HgbA1c. | 3 months
To determine if the addition of sitagliptin changes tacrolimus or sirolimus drug levels in post-kidney transplant patients | 3 months
Determine tolerability of sitagliptin therapy in post-kidney transplant patients. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James T Lane, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States